CLINICAL TRIAL: NCT02508103
Title: Emotional Processing and Oxytocin Mechanisms in Premenstrual Dysphoric Disorder: A Pilot Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Susan Girdler, PhD, Principal Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14-1153
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Premenstrual Dysphoric Disorder
Keywords: Premenstrual Dysphoric Disorder; Premenstrual Syndrome; PMS; PMDD
MeSH Terms: conditions — Premenstrual Dysphoric Disorder; Premenstrual Syndrome | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin, then Placebo (Experimental): Participants were randomized to receive Intransal Oxytocin for late luteal phase administration during one menstrual cycle, then received Intranasal Placebo for late luteal phase administration of a subsequent menstrual cycle.
  Intranasal Oxytocin spray (40 IU, 3x/day) for 4-5 days; Intranasal Placebo spray (3x/day) for 4-5 days
  Interventions: Drug: Oxytocin; Drug: Placebo
- Placebo, then Oxytocin (Experimental): Participants were randomized to receive Intranasal Placebo for late luteal phase administration during one menstrual cycle, then received Intransal Oxytocin for late luteal phase administration of a subsequent menstrual cycle.
  Intranasal Oxytocin spray (40 IU, 3x/day) for 4-5 days; Intranasal Placebo spray (3x/day) for 4-5 days
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Intranasal Oxytocin spray (40 IU, 3x/day) self-administered during laboratory testing session and then for 4-5 days until menses begins
Drug: Placebo — Intranasal Placebo spray (3x/day) self-administered during laboratory testing session and then for 4-5 days until menses begins

SUMMARY:
This research study will look at brain and symptom differences among women with severe premenstrual mood symptoms. One goal of this study is to look at the effects of taking a nasal spray containing oxytocin (a hormone made in the brain) on brain areas involved in emotion regulation while viewing pictures during a neuroimaging (fMRI) session. The investigators will also look at whether oxytocin improves premenstrual mood symptoms.

DETAILED DESCRIPTION:
Purpose: The primary objective of this pilot study is to use functional neuroimaging techniques to begin to identify the central brain networks that may contribute to impairment in emotion regulation, interpersonal relationships, and marital and family function in women with premenstrual dysphoric disorder (PMDD), particularly for those women who also have a history of early life abuse (ELA).

Based on the evidence that the mammalian neuropeptide oxytocin (OT), best known for its role in lactation and parturition, plays a seminal role in social affiliation, emotion regulation, attachment, maternal behavior, trust, and protection against stress; and because OT neural pathways and receptors are prominently expressed in brain regions involved in emotion regulation and maternal/affiliative behavior; the study will: 1) use intranasal OT administration as a probe to assess whether it modifies activation of brain regions involved in emotion regulation in response to an emotional processing task; and 2) whether daily intranasal OT administration during the premenstrual phase improves symptoms in women with PMDD with or without a history of ELA.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to enter this study, subjects will have met PMDD Study Entry Criteria in the diagnostic feeder study (IRB# 05-3000)
* 18 to 52 years of age
* Regular menstrual cycles
* Ability to give informed consent

Exclusion Criteria:

* current psychiatric diagnosis of substance abuse or claustrophobia (fear of closed places)
* pregnancy (based on urine pregnancy test) or breastfeeding
* use of psychiatric medication (e.g. for depression, anxiety), hormonal medication, other agents that alter mood or thinking, or street drugs
* any foreign iron or steel metal objects in the body, such as a pacemaker, shrapnel, metal plate, certain types of tattoos, or metal debris

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Girdler, PH.D., Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxytocin, Then Placebo: Participants were randomized to receive Intransal Oxytocin for late luteal phase administration during one menstrual cycle, then received Placebo for late luteal phase administration of a subsequent menstrual cycle.
  Intranasal Oxytocin spray (40 IU, 3x/day) for 4-5 days; Intranasal Placebo spray (3x/day) for 4-5 days
- Placebo, Then Oxytocin: Participants were randomized to receive Intransal Placebo for late luteal phase administration during one menstrual cycle, then received Oxytocin for late luteal phase administration of a subsequent menstrual cycle.
  Intranasal Oxytocin spray (40 IU, 3x/day) for 4-5 days; Intranasal Placebo spray (3x/day) for 4-5 days
Period: Overall Study
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Within-person experimental design, each participant received oxytocin and placebo.
Groups:
- Placebo, Then Oxytocin: Participants were randomized to receive Intransal Placebo for late luteal phase administration during one menstrual cycle, then received Intranasal Oxytocin for late luteal phase administration of a subsequent menstrual cycle.
  Intranasal Oxytocin spray (40 IU, 3x/day) for 4-5 days; Intranasal Placebo spray (3x/day) for 4-5 days
- Total: Total of all reporting groups
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 36.4 [28 to 45] | 36.8 [31 to 41] | 36.6 [28 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Premenstrual Symptom Severity
Description: The investigators will analyze premenstrual symptom severity ratings during the late luteal phase of two consecutive menstrual cycles to assess the effects of intranasal oxytocin (vs. placebo) on premenstrual symptom severity. Daily premenstrual symptoms were measured using the Daily Record of Severity of Problems (DRSP; Endicott et al., 2006). Across 24 items representing emotional, physical, and behavioral symptoms, participants indicated "the degree to which the problems have been experienced today": 1-Not at all, 2-Minimal, 3-Mild, 4-Moderate, 5-Severe, or 6-Extreme. For each participant, we calculated a total score by summing all 24 items. We then calculated a mean total score for each condition by averaging all participants total scores in a given condition. Higher scores represent greater symptoms. Range of total score is 24 to 144.
Time Frame: During the late luteal phase of two consecutive menstrual cycles (an average of 3-5 days of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Oxytocin: Intranasal Oxytocin spray (40 IU, 3x/day) for 4-5 days
- Placebo: Intranasal Placebo spray (3x/day) for 4-5 days
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | 25.05 (16.74) | 27.36 (13.80)

2. Primary Outcome: Amygdala Response to Cognitive-emotional Processing Task During Functional Magnetic Resonance Imaging (fMRI)
Description: During fMRI scanning, the investigators will assess the effects of intranasal oxytocin (vs. placebo) on amygdala response to cognitive-emotional processing task (Hariri et al., 2006) during the late luteal phase of two consecutive menstrual cycles. Amygdala reactivity was assessed by extracting a "contrast of parameter estimate" (COPE) for each region (left and right amygdala). Regions were defined using binarized Harvard-Oxford Subcortical Atlas masks. The parameter estimate was the average estimate of all voxels in each region for the task contrast of viewing Faces vs. Shapes. We used neuroimaging software package FSL to calculate and extract these parameter estimates.
Time Frame: 1 hour of scanning during the late luteal phase of two consecutive menstrual cycles
Measure: Mean (Standard Deviation); unit: parameter estimate
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 10 | 10
parameter estimate
  Left Amygdala | 0.89 (0.48) | 0.95 (0.81)
  Right Amygdala | 1.14 (0.57) | 1.22 (1.25)

ADVERSE EVENTS:
Time Frame: Systematic assessment of adverse events occurred during intranasal oxytocin and placebo administration; each assessment occurred on the 3rd day of at-home administration. Participants were asked to report any other adverse events throughout their enrollment in the study (minimally: 2 months, maximally: 5mos).
Description: For systematic assessment of adverse events during administration of nasal sprays, we reviewed various symptoms with participants over the phone; response options for each symptom were "yes/no". If participants endorsed a symptom (e.g., headache), we collected information on severity, whether or not it might be related to the study, whether the symptom resolved, and whether the symptom led to drop out.
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=10) | Placebo (N=10)
Headache (Nervous system disorders) | 2 (2) | 0 (0) — Mild headache reported by two participants during oxytocin administration.
Uterine cramps (Reproductive system and breast disorders) | 2 (2) | 0 (0) — Mild uterine cramping reported by two participants during oxytocin administration.
Clogged nostril (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Participant reported one nostril became slightly clogged during intranasal Placebo administration.

LIMITATIONS AND CAVEATS:
Results of this study should be interpreted with caution due to the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes